CLINICAL TRIAL: NCT00394888
Title: Hemangioma Associated With High Rates of Morbidity:A Prospective Study
Brief Title: Hemangioma Associated With High Rates of Morbidity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: University of California, San Francisco (Other); Columbia University (Other); Baylor College of Medicine (Other); St. Justine's Hospital (Other); State University of New York - Downstate Medical Center (Other); Children's Mercy Hospital Kansas City (Other); Children's Hospital Medical Center, Cincinnati (Other); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Principal Investigator, Beth Drolet, Professor and Vice Chair of Dermatology, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: High Risk Hemangioma
Record Dates: First submitted 2006-11-01; First posted 2006-11-02 (Estimated); Results first posted 2011-07-06 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Hemangioma
Keywords: Hemangioma; PHACE; Lumbosacral hemangioma; Occult Spinal Dysraphism
MeSH Terms: conditions — Hemangioma; Neural Tube Defects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Facial Hemangioma (Other): Patients with large facial hemangioma.
  Interventions: Device: MRI of head and neck; Other: Dermatological Examination; Other: Cardiac examination
- Lumbosacral Hemangioma (Other): Patients with lumbosacral hemangioma.
  Interventions: Device: MRI; Other: Dermatological Examination
- Multiple Hemangiomas (Other): patients with multiple hemangiomas (>5)
  Interventions: Device: MRI; Other: Dermatological Examination; Device: Abdominal ultrasound

INTERVENTIONS:
Device: MRI — MRI of the spine.
  Arms: Lumbosacral Hemangioma; Multiple Hemangiomas
Device: MRI of head and neck — MRI of head and C-spine
  Arms: Facial Hemangioma
Other: Dermatological Examination — Complete dermatological examination to identify and characterize nature of dermatological anomalies
  Other Names: Clinical dermatological examination
Other: Cardiac examination — Complete cardiac examination
  Other Names: Cardiovascular examination
  Arms: Facial Hemangioma
Device: Abdominal ultrasound — Abdominal ultrasound to detect hepatic hemangiomas
  Arms: Multiple Hemangiomas

SUMMARY:
We are conducting a study on the possible presence of PHACES in children with large facial hemangiomas and lumbosacral hemangiomas of infancy (hemangioma in the lower back) . With this study we hope to better understand the risk of this syndrome and to develop guidelines for its evaluation and management.

DETAILED DESCRIPTION:
Large hemangiomas of the face can be associated with anomalies of the blood vessels of head and chest. The acronym PHACES indicates the association of Posterior fossa and other brain malformations, facial Hemangioma, Arterial anomalies, Coarctation of the aorta and other cardiac defects, Eye abnormalities and Sternal malformations. Study subjects will be recruited through the Pediatric Dermatology department in several cities. All patients age 0-1 year old of age, who present with large facial hemangioma (>22 cm^2) will be offered to participate in the study. Parents will be interviewed to obtain personal, medical, and family history.

Patients will undergo standard of care evaluation for facial hemangioma with risk of PHACE syndrome. This includes skin, eye and neurological examination, photograph, magnetic resonance imaging (MRI) of head/neck/chest, and lab tests requiring samples of blood, urine or stool. No other tests will be performed for participating in the study.

Lumbosacral hemangiomas of infancy (hemangioma in the lower back) can be associated with anomalies of the spine. "Tethered cord syndrome" indicates a condition caused by abnormally stretched spinal cord. Over time this condition can lead to neurological damage. Although often there are no symptoms until adulthood, it can become apparent during childhood. Common symptoms are: lower back pain, pain and weakness of the legs, walking problems, and bladder and bowel loss of control. "Occult spinal dysraphism" is the term used when the defect of the spine is hidden under normal skin. We noticed that infants with hemangioma in the lower back area are more inclined to present a hidden spine defect.

Study subjects will be recruited through the Pediatric Dermatology departments in several cities. All patients age 0-18 year old of age, who present with lumbosacral hemangioma (> 2.5 cm of diameter overlying the spine) will be offered to participate in the study. Parents will be interviewed to obtain personal, medical, and family history.

Patients will undergo standard of care evaluation for lumbosacral hemangioma. This includes skin, neurological examination, photograph, magnetic resonance imaging (MRI) of the back, lab tests requiring samples of blood, urine or stool. No additional tests will be performed only for participating in the study.

ELIGIBILITY:
Segmental Facial Hemangioma

Inclusion criteria:

* Infants less than 1 year of age
* Hemangiomas of the head /facial area measuring 22cm2 or greater.

Exclusion criteria:

* Children greater than 1 year of age.
* Children with segmental hemangiomas present in locations other than the head.
* Children presenting with localized (focal) or indeterminate hemangiomas in any location.
* Children with other vascular tumors (such as tufted angioma, Kaposiform hemangioendothelioma, non-involuting congenital hemangioma or rapidly-involuting congenital hemangioma) or vascular malformations.

Lumbosacral Hemangioma

Inclusion criteria:

* Individuals less than 18 years of age.
* Hemangioma, hemangioma precursor, or definitive residual hemangioma larger then 2.5 cm in diameter, overlying the midline lumbar spine or sacral spine in which any portion of the hemangioma is located over the midline.

Exclusion Criteria:

* Excluding perirectal hemangiomas that do not extend onto the sacral spine.
* Excluding perineal hemangiomas that do extend to overlay the sacral spine.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 433 (Actual)
Dates: Start 2005-11; Primary Completion 2009-11 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth Drolet, MD, Principal Investigator — Medical College of Wisconsin; Maria Garzon, MD, Principal Investigator — Columbia University; Denise Metry, MD, Principal Investigator — Baylor College of Medicine; Ilona Frieden, MD, Principal Investigator — University of California, San Francisco; Julie Powell, MD, Principal Investigator — Hopital Sainte-Justine; Anne Lucky, MD, Principal Investigator — Children's Hospital of Cincinnati; Sharon Glick, MD, Principal Investigator — State University of New York - Downstate Medical Center; Eulalia Baselga, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Anita Haggstrom, M.D., Principal Investigator — Indiana University; Anthony Mancini, MD, Principal Investigator — Northwestern University; Kimberly Horii, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Beth Drolet, MD, Milwaukee, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Multiple Hemangiomas: Patients with multiple hemangiomas
Period: Overall Study
Arm/Group | Facial Hemangioma | Lumbosacral Hemangioma | Multiple Hemangiomas
Started | 108 | 48 | 201
Completed | 108 | 48 | 201
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Facial Hemangioma | Lumbosacral Hemangioma | Multiple Hemangiomas | Total
Number analyzed (Participants) | 108 | 48 | 201 | 357
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 108 | 48 | 201 | 357
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 0.5 (1) | 0.5 (1) | 0.5 (1) | 0.5 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 33 | 152 | 263
  Male | 30 | 15 | 49 | 94
Region of Enrollment [Number; unit: participants]
  United States | 108 | 48 | 201 | 357

OUTCOME MEASURES:

1. Primary Outcome: MRI/MRA of Head/Neck/Chest.
Time Frame: 2 years
Measure: Number; unit: participants
Groups:
- All Participants: entire population count for MRI/A
Arm/Group | All Participants
Number analyzed (Participants) | 357
participants | 357

2. Primary Outcome: Clinical Diagnosis of PHACE Syndrome
Description: For subjects in the large facial hemangioma arm of the study, a clinical assessment by trained physicians was conducted to determine whether or not each subject met diagnostic criteria for PHACE syndrome.
Time Frame: 2 years
Population: Subjects enrolled in the large facial hemangioma arm (n= 108) were analyzed for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 108
Participants | 33

3. Primary Outcome: Spinal Abnormalities
Description: The number of lumbrosacral hemangioma subjects with confirmed spinal abnormalities detected via lumbrosacral MRI.
Time Frame: 2 years
Population: Subjects enrolled in the lumbrosacral hemangioma arm (n= 48) were analyzed for this outcome measure
Measure: Number; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 48
Participants | 21

4. Primary Outcome: Cerebrovascular and Structural Brain Abnormalities
Description: The number of PHACE subjects identified with cerebrovascular and/or structural brain abnormalities detected using MRI.
Time Frame: 2 years
Population: Subjects diagnosed with clinically definite PHACE syndrome, enrolled in the large facial hemangioma arm (n= 33) were analyzed for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 33
Participants | 31

5. Primary Outcome: Cardiac Abnormalities Detected Via Clinical Examination
Description: The number of subjects with clinically definite PHACE syndrome who were identified as having cardiac abnormalities following clinical examination.
Time Frame: 2 years
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 33
Participants | 22

6. Primary Outcome: Frequency of Hepatic Hemangiomas Detected Via Abdominal Ultrasound
Description: The number of participants with multiple (greater than or equal to 5) cutaneous infantile hemangiomas who were found to have hepatic hemangiomas via the us abdominal ultrasound.
Time Frame: 2 years
Population: Subjects enrolled in the hepatic hemangioma arm (n= 151) were analyzed for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 151
Participants | 24

ADVERSE EVENTS:
Arm/Group | Facial Hemangioma | Lumbosacral Hemangioma | Multiple Hemangiomas
Serious Adverse Events (participants affected / at risk) | 0/108 | 0/48 | 0/201
Other Adverse Events (participants affected / at risk) | 0/108 | 0/48 | 0/201

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes